CLINICAL TRIAL: NCT00763152
Title: The Probe Study - The PROstate Bed Evaluation - A Study to Record the Implant Experience, Transponder Stability and Tracking Data of the Calypso 4D Localization Study in the Prostate Bed
Brief Title: CMT-07-08: The PROstate Bed Evaluation Study
Status: Completed | Type: Observational
Sponsor: Varian, a Siemens Healthineers Company (Industry)
Responsible Party: Sponsor
Other Study IDs: CMT-07-08
Record Dates: First submitted 2008-09-25; First posted 2008-09-30 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: prostate; prostate bed; periprostatic
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- stability of Beacons in prostatic bed: Patients implanted with the Calypso transponders following radical prostatectomy for prostate cancer will be followed for observation of transponder stability.
  Interventions: Other: Observation of transponder stability

INTERVENTIONS:
Other: Observation of transponder stability — Observation of transponder stability and placement in the prostatic bed following radical prostatectomy

SUMMARY:
This is an observational study to collect placement and tracking data for patients who have the Calypso transponders implanted into the peri-prostatic tissue.

DETAILED DESCRIPTION:
Use of Real-time tracking using Calypso Electromagnetic Beacons in the prostatic bed of patients receiving radiotherapy following radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrence of prostate cancer following radical prostatectomy for prostate adenocarcinoma
2. Patients with initially undetectable PSA following prostatectomy for prostate adenocarcinoma with subsequent PSA relapse
3. Patients being planned for radiation therapy
4. Patient is being planned for implant with Calypso Transponders in the prostate bed
5. No evidence of distant metastases
6. Age ≥ 18 years
7. Informed consent

Exclusion Criteria:

1. The patient has received other investigational therapy in the last 60 days
2. The patient has previously been implanted with permanent beacon transponders
3. The patient has a prosthetic implant in the pelvic region that contain metal or conductive materials
4. The patient has any other medical or other condition that would, in the investigator's opinion, make them a poor candidate for the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer of the peri-prostatic tissue or prostate bed
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2008-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
To collect data on the process of implanting the Calypso Transponder in the prostate bed following radical prostatectomy | Immediate

SECONDARY OUTCOMES:
Evaluate the stability of the Calypso transponder in the prostate bed | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Rajanish Singla, MD, Principal Investigator — Metro Uro-Rad
Locations (2):
- United States (2):
  - 21C Oncology - Scottsdale, Scottsdale, Arizona
  - Metropolitan Uro-Rad, St Louis, Missouri

REFERENCES:
- [Background] Balter JM, Wright JN, Newell LJ, Friemel B, Dimmer S, Cheng Y, Wong J, Vertatschitsch E, Mate TP. Accuracy of a wireless localization system for radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Mar 1;61(3):933-7. doi: 10.1016/j.ijrobp.2004.11.009. PMID 15708277
- [Background] Litzenberg DW, Willoughby TR, Balter JM, Sandler HM, Wei J, Kupelian PA, Cunningham AA, Bock A, Aubin M, Roach M 3rd, Shinohara K, Pouliot J. Positional stability of electromagnetic transponders used for prostate localization and continuous, real-time tracking. Int J Radiat Oncol Biol Phys. 2007 Jul 15;68(4):1199-206. doi: 10.1016/j.ijrobp.2007.03.030. Epub 2007 May 21. PMID 17513060
- [Background] Kupelian P, Willoughby T, Mahadevan A, Djemil T, Weinstein G, Jani S, Enke C, Solberg T, Flores N, Liu D, Beyer D, Levine L. Multi-institutional clinical experience with the Calypso System in localization and continuous, real-time monitoring of the prostate gland during external radiotherapy. Int J Radiat Oncol Biol Phys. 2007 Mar 15;67(4):1088-98. doi: 10.1016/j.ijrobp.2006.10.026. Epub 2006 Dec 21. PMID 17187940